CLINICAL TRIAL: NCT06472310
Title: An Observational Multicenter Cross-sectional Study of Patients With Uncontrolled Severe Asthma in the Population of the Russian Federation
Brief Title: Clinical and demOgRaphic Features of Patients With Uncontrolled Severe Asthma in Russia (CORSAR)
Acronym: CORSAR
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5180R00037
Record Dates: First submitted 2024-05-22; First posted 2024-06-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Severe Asthma
Keywords: uncontrolled severe asthma; SA
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is an observational multicenter cross-sectional study. Planned study population consists of 5 000 adult patients with uncontrolled SA receiving treatment according to standard of care (except biologics). Planned number of study site is 50 outpatient centers with experience of uncontrolled SA treatment in about 50 regions of Russia (in order to describe characteristics of patients with uncontrolled SA in different regions in the most comprehensive way). This non-interventional study does not imply any intervention into a routine clinical practice, and does not provide for any diagnostic and therapeutic procedures other than those used in routine practice.

DETAILED DESCRIPTION:
There are limited epidemiological data of the patients with uncontrolled severe asthma in Russia since there is no unified system for regular monitoring of patients with severe asthma in the country. The systematic information about complications and comorbidities, about the treatment approaches and their effectiveness in the Russian population is also absent.

The observational registry is really important to describe the epidemiological characteristics of the disease and to analyse the clinical characteristics of the various subgroups of patients. This is an excellent starting point to be able to investigate the characteristics of the disease in detail.

The Russian Federation consists of 85 regions with a total population of more than 145 million people. The regions differ in ethnic composition, age, gender, climate, ecology, economic level, prevalence of asthma in general and severe asthma in particular.

Previously reported observational registries are International Severe Asthma Registry (ISAR) and Russian Severe Asthma Registry (RSAR), both studies included patients regardless of whether patients received biological agents or not. The percentage of patients receiving biologics in these studies was 25.4% and 10.6% respectively.

Thus, there is a need to perform a large-scale observational registry in regions of the country with a sufficient size of population to obtain information on SA epidemiology, clinical and demographic characteristics, to describe main clinical outcomes and evaluate existing associations between observed treatment patterns and clinical outcomes in real clinical practice in patients with uncontrolled SA not receiving biologic therapy.

Trial will have cross-sectional design and will include 1 visit for obtaining the patient's demographic and clinical data. To allow wide data coverage the study will involve at least 50 regions of Russian Federation; in each region 100 patients will be recruited. The total size of study population will be 5 000 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of inclusion;
2. Signed and dated written informed consent in accordance with ICH GCP and local law prior to inclusion in the study;
3. Patients with diagnosis of uncontrolled SA (Asthma Control Questionnaire-5 (ACQ-5) score > 1,5) established no less than 52 weeks prior to inclusion; Severe asthma is defined as asthma, that is controlled due to treatment with ICS in medium or high doses plus LABA and/or ALP, and/or LAMA, and/or systemic corticosteroids (sCS), and/or immunobiological therapy, while attempts to reduce the volume of therapy lead to a loss of symptom control, or asthma remains uncontrolled despite this treatment. Such therapy should be carried out at least 3 months before inclusion.

   Uncontrolled asthma is defined as ACQ-5>1.5.
4. Patients with the availability of at least 52 weeks of follow-up data (prior to inclusion) in the medical records.

Exclusion Criteria:

1. Patients receiving any biological therapy currently or within 52 weeks prior to inclusion;
2. Presence of chronic obstructive pulmonary disease (COPD) or idiopathic pulmonary fibrosis (ILF) currently or in the anamnesis;
3. The participation in any clinical study currently or within 52 weeks prior to inclusion;
4. An acute or chronic disease that, as deemed by Investigator, limits the ability of patients to participate in this study or could influence the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 5 000 adult patients with confirmed diagnosis of uncontrolled SA who receive medical treatment (excluding biological therapy) and are monitored and treated by pulmonologists or allergologists in approximately 50 clinical centers in about 50 regions of Russia
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
To characterise the profile of routine therapy used for patients with uncontrolled SA not receiving biological therapy in proportion of patients receiving different classes of drugs will be calculated | June 2024 - June 2027
  1. ICS alone (duration, dosage);
  2. LABA alone (duration, dosage);
  3. ICS and LABA (duration, dosage);
  4. ICS and LABA plus:
  a. Short-acting beta-agonists (SABA) (duration, dosage); b. LAMA (duration, dosage); c. LTRA (duration, dosage); d. Theophylline (duration, dosage); e. Macrolide antibiotics (duration, dosage).
To determine the pattern and trends of OCS prescription | June 2024 - June 2027
  Proportion of patients receiving OCS: intermittent/regularly; Median daily dose in case of regular OCS use; Median cumulative OCS exposure.
To describe clinical and demographic characteristics of patients with uncontrolled SA not receiving biological therapy in Russian Federation mean age at the inclusion into the study will be collected | June 2024 - June 2027
To describe demographic characteristics of patients with uncontrolled SA not receiving biological therapy in Russian Federation mean age at the primary asthma diagnosis will be collected | June 2024 - June 2027
To describe demographic characteristics of patients with uncontrolled SA not receiving biological therapy in Russian Federation mean age at the diagnosis of SA will be collected | June 2024 - June 2027
To describe demographic characteristics of patients with uncontrolled SA not receiving biological therapy in Russian Federation proportion of men and women will be calculated | June 2024 - June 2027
To describe demographic characteristics of patients with uncontrolled SA not receiving biological therapy in Russian Federation data on mean body mass index (BMI) will be collected | June 2024 - June 2027
To describe demographic characteristics of patients with uncontrolled SA not receiving biological therapy in Russian Federation proportion of patients with overweight will be calculated | June 2024 - June 2027
  BMI ≥25 kg/m2
To describe demographic characteristics of patients with uncontrolled SA not receiving biological therapy in Russian Federation data on proportion of patients with different educational statuses | June 2024 - June 2027
  educational statuses: higher, secondary special, secondary general
To describe demographic characteristics of patients with uncontrolled SA not receiving biological therapy in proportion of patients from each residential region of Russia will be calculated | June 2024 - June 2027
To describe demographic characteristics of patients with uncontrolled SA not receiving biological therapy in Russian Federation proportion of patients with negative lifestyle factors will be calculated | June 2024 - June 2027
  1. Proportion of patients with history of smoking/current smokers;
  2. Mean smoking index (pack-years) for current smokers;
  3. Proportion of patients with a history of alcohol abuse/current alcohol abuse;
  4. Proportion of patients with limitation of physical activity, related/non-related to asthma;
  5. Proportion of patients with overweight (BMI ≥25 kg/m2).
To describe clinical characteristics of patients with uncontrolled SA not receiving biological therapy in Russian Federation proportion of patients with chronic rhinosinusitis with nasal polyps will be calculated | June 2024 - June 2027
  Proportion of patients with chronic rhinosinusitis with nasal polyps (CRSwNP), overall proportion and:
  a. Proportions of patients with CRSwNP with different levels of eosinophils blood count: i. <150 cells/μl; ii. ≥150 cells/μl; iii. ≥300 cells/μl. b. Proportions of patients with CRSwNP with different levels of total IgE: i. ≤30 UI/ml; ii. >30 UI/ml; c. The proportion of patients with CRSwNP with a history of prior biologic treatment ('any biologic drugs used for asthma treatment in the past'); d. The proportion of patients with CRSwNP who were recommended to start biologic treatment at the first visit ('the need of biological therapy prescription').
To describe clinical characteristics of patients with uncontrolled SA not receiving biological therapy in Russian Federation proportion of patients with different comorbidities will be calculated | June 2024 - June 2027
To describe clinical characteristics of patients with uncontrolled SA not receiving biological therapy in Russian Federation mean eosinophils blood count will be collected | June 2024 - June 2027
  cells/μl
To describe clinical characteristics of patients with uncontrolled SA not receiving biological therapy in Russian Federation proportion of patients with different levels of eosinophils blood count will be calculated | June 2024 - June 2027
  1. <150 cells/μl;
  2. ≥150 cells/μl;
  3. ≥300 cells/μl.
To describe clinical characteristics of patients with uncontrolled SA not receiving biological therapy in Russian Federation 14. Mean eosinophils count in sputum will be collected | June 2024 - June 2027
  cells per high power field
To describe clinical characteristics of patients with uncontrolled SA not receiving biological therapy in Russian Federation 15. Mean total Immunoglobulin E will be calculated | June 2024- June 2027
  IU/ml
To describe clinical characteristics of patients with uncontrolled SA not receiving biological therapy in Russian Federation proportion of patients with different levels of total IgE will be calculated | June 2024 - June 2027
  1. ≤30 UI/ml;
  2. >30 UI/ml;
To describe clinical characteristics of patients with uncontrolled SA not receiving biological therapy in Russian Federation mean FeNO will be calculated | June 2024 - June 2027
  parts per billion (ppb)

SECONDARY OUTCOMES:
1. Proportion of patients with change of inhaled therapy during retrospective 52-week follow-up period | June 2024 - June 2027
  1. Change of ICS;
  2. Dose of ICS increased;
  3. Addition of another drug for inhaled therapy
2. Proportion of patients with OCS prescription occurred during retrospective 52-week follow-up period | June 2024 - June 2027
3. Proportion of participants sent to biological therapy | June 2024 - June 2027
4. Proportion of patients experiencing 0, 1, 2, ≥3 severe asthma exacerbations* during retrospective 52-week follow-up period | June 2024 - June 2027
  *Severe asthma exacerbation is defined as worsening of asthma requiring any of the following:
  * use of systemic corticosteroids (CS) (or a temporary increase in a stable OCS background dose) for at least 3 days or a single depo-injectable dose of CS and/or
  * an emergency room/urgent care visit (defined as evaluation and treatment for < 24 hours in an emergency department or urgent care center) due to asthma that required systemic CS (as per above) and/or
  * an inpatient hospitalization (defined as admission to an inpatient facility and/or evaluation and treatment in a healthcare facility for ≥ 24 hours) due to asthma.
5. Annualised rate of severe asthma exacerbations* during retrospective 52-week follow-up period | June 2024 - June 2027
6. Cumulative days of severe asthma exacerbations | June 2024 - June 2027
7. Proportion of patients with healthcare resource utilization (HRU) events during retrospective 52-week follow-up period: | June 2024 - June 2027
  1. Unscheduled outpatient visits;
  2. Emergency department visits/emergency calls;
  3. Hospitalizations.
8. Mean parameters of lung function: | June 2024 - June 2027
  1. Mean pre- and post-bronchodilator forced expiratory volume in 1 second (pre- and post-FEV1);
  2. Mean pre- and post-bronchodilator forced vital capacity (pre- and post-FVC);
  3. Mean pre-bronchodilator forced expiratory flow (pre-FEF);
  4. Mean functional residual capacity (FRC), residual lung volume (RLV) and total lung capacity (TLC) evaluated by spirometry and/or body plethysmography.

CONTACTS AND LOCATIONS:
Locations (38):
- Russia (38):
  - Research Site, Astrakhan
  - Research Site, Barnaul
  - Research Site, Blagoveshchensk
  - Research Site, Bryansk
  - Research Site, Chelyabinsk
  - Research Site, Gatchina
  - Research Site, Irkutsk
  - Research Site, Izhevsk
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Khabarovsk
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Murmansk
  - Research Site, Nal'chik
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Orenburg
  - Research Site, Petrozavodsk
  - Research Site, Rostov-on-Don
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Saratov
  - Research Site, Smolensk
  - Research Site, Stavropol
  - Research Site, Tomsk
  - Research Site, Ufa
  - Research Site, Ulan-Ude
  - Research Site, Verkhnyaya Pyshma
  - Research Site, Vladimir
  - Research Site, Vladivostok
  - Research Site, Volgograd
  - Research Site, Voronezh
  - Research Site, Yakutsk
  - Research Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/